CLINICAL TRIAL: NCT04529382
Title: Neurodevelopmental Outcome After Fetal Neonatal AlloImmune Thrombocytopenia
Acronym: NOFNAIT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Leiden University Medical Center (Other)
Collaborators: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Responsible Party: Principal Investigator, elopriore, Prof. E. Lopriore, Leiden University Medical Center
Other Study IDs: P19.069
Record Dates: First submitted 2020-07-15; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Fetal and Neonatal Alloimmune Thrombocytopenia; Long Term Adverse Effects; Neurodevelopmental Abnormality; Intravenous Immunoglobulin Adverse Reaction
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune; Long Term Adverse Effects | interventions — Neurologic Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Unanticipated FNAIT cases: All children born between 2002 and 2017 and diagnosed with FNAIT are eligible for this study. Children in cohort 1 will be FNAIT cases that were not antenatally treated with by maternal IVIg administration (or other forms of fetal therapy).
  Interventions: Diagnostic Test: Cognitive testing (Bayley III, WPPSI III and WISC V)
- Cohort 2: Anticipated FNAIT cases: All children born between 2002 and 2017 and diagnosed with FNAIT are eligible for this study. Children in cohort 2 will be FNAIT cases which were anticipated antenatally by maternal IVIg administration according to our local protocol.
  Interventions: Diagnostic Test: Cognitive testing (Bayley III, WPPSI III and WISC V)

INTERVENTIONS:
Diagnostic Test: Cognitive testing (Bayley III, WPPSI III and WISC V) — Parents and children will be invited to come for an outpatient clinic visit where cognitive testing and neurologic examination will be performed. In addition to this parents will be asked to fill in questionnaires, provide latest school results and medical files will be requested from treating physicians.
  Other Names: Pediatric Quality of Life Inventory; Child Behavior Checklist; Questionnaire based on 'Richtlijn diagnostiek naar onderliggende aandoeningen bij kinderen met recidiverende luchtweginfecties'; Questionnaire composited in collaboration with allergist (Dr. H. de Groot).; Neurologic Examination

SUMMARY:
Fetal and neonatal alloimmune thrombocytopenia (FNAIT) is a disease caused by allo-immunisation during pregnancy. If left untreated, FNAIT can lead to severe fetal intracranial haemorrhage. This complication can be prevented by weekly administration of intravenous immunoglobulin (IVIg) to the mother during pregnancy. Knowledge on long-term development of FNAIT survivors with or without IVIg treatment is very limited but an important subject in the counselling of parents of newly diagnosed cases. To evaluate the long-term neurodevelopmental outcome in two groups of children with FNAIT will be asked to participate in our study in an outpatient clinic setting.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Fetal and neonatal alloimmune thrombocytopenia (FNAIT) is the most common cause of thrombocytopenia in otherwise healthy term-born neonates. FNAIT is a rare disease with an incidence estimated around 1 per 1000 live newborns. During pregnancy alloimmunization can occur due to incompatibility of the Human Platelet Antigens (HPA) on the maternal and fetal platelets. Alloimmunization and maternal production of antibodies directed against the HPA-positive fetal platelets, leads to thrombocytopenia and an increased risk of intracranial hemorrhages (ICH) in the fetus. Clinical presentation can vary from skin bleedings to severe ICH leading to lifelong neurologic sequelae or intrauterine death.

In the past, FNAIT was managed with invasive and high-risk interventions including intrauterine platelet transfusion (IUPT). Since the end of the 20th century, invasive intrauterine transfusions (IUT) were replaced by a new, non-invasive therapy: maternal administration of intravenous immunoglobulin (IVIg). This novel therapy resulted in a significant lower risk of intrauterine fetal death and ICH. Intervention with immune modulation in the semi -allogenic environment of the fetus by administration of immunoglobulins (Ig) is successful, especially in preventing ICH. However antenatal treatment with IVIg has been implemented as standard of care without strong methodological follow-up research of children from mothers treated with IVIg. To date, only two follow-up studies have been published in children with anticipated FNAIT cases. The first study of a FNAIT cohort treated with IVIg was done by Ward et al. in 2006. They concluded that development of children treated for FNAIT was better compared to their non-treated siblings. Their conclusions were based on non-validated questionnaires taken by telephone, assessing the behavioral outcome of the children and were limited by a ~40% lost-to-follow-up rate. A second follow-up study including 39 children was published by a research group from our center in 2004. This research stated that the outcome in children with FNAIT and exposed to maternal IVIg treatment was similar to the normal population. However, this study included a heterogenic group of children with different treatment strategies including IUT, hampering definitive conclusions and substantiating the need for more research.

No long-term standardized follow-up studies were performed on FNAIT cases without antenatal treatment and/or ICH. The natural course of the disease and long-term effects of thrombocytopenia on the developing fetus and newborn are unknown. FNAIT is defined as a disease caused by alloantibodies, resulting in thrombocytopenia and a risk of bleeding in the neonate. In the last years, evidence is increasing that the maternal alloantibodies can also bind to the fetal endothelium and may impair angiogenesis in the developing fetuses It is not known at which moment in pregnancy the developing brain is most vulnerable for damage induced by these kind of alloantibodies. The timing in fetal life FNAIT associated ICH ranges from 23 to 42 weeks, but small bleeding may not be diagnosed. It may also be that these type of alloantibodies not lead to ICH but to other type of cerebral damage. These lesions can remain subclinical directly after birth but lead to developmental delay on the long term. This knowledge can be of great interest when counseling parents with a risk of FNAIT or in writing guidelines.

For 3 decades a nationwide screening on FNAIT to detect pregnancies with alloantibodies in time and start treatment to prevent bleedings is being discussed. If alloantibodies lead to cerebral damage on the long term also in patients without large ICH this might have large implications in the debate on the introduction of a national screening programme. Therefore the investigators want to underline that more knowledge about the long-term development of FNAIT survivors is required.

The Leiden University Medical Center (LUMC), a national fetal therapy center in The Netherlands, has a close and long-lasting collaboration with Sanquin. This collaboration offers a unique opportunity to evaluate a large and complete cohort of children with FNAIT. LUMC and Sanquin are both nationwide referral centers for FNAIT and committed to improve timely detection of high-risk cases who need intra-uterine therapy. This research group from the national expertise centers are designated to assess long-term outcome in children with FNAIT and describe the natural history of children affected by FNAIT and the long term effects of a given therapy.

OBJECTIVE The primary objective is to determine the cognitive test score of children diagnosed with FNAIT without and with antenatal treatment.

STUDY DESIGN The investigators will perform an observational cohort study. The long-term neurodevelopmental outcome of children affected by FNAIT will be evaluated. All children born between 2002 and 2017 and diagnosed with FNAIT are eligible for follow-up assessment and will be invited for an assessment at our outpatient clinic. The FNAIT survivors will be collected in two cohorts; cohort 1 will consist of FNAIT survivors without antenatal treatment, cohort 2 will consist of FNAIT survivors that were antenatally anticipated and therefore IVIg treatment to the mother was given.

Enrollment in this study will take place via the LUMC and Stichting Sanquin Bloedvoorziening. The LUMC is national referral center for intrauterine therapy and Sanquin is national reference laboratory to diagnose FNAIT. Retrospectively FNAIT cases will be collected and asked for permission directly or via referring specialist.

After informed consent, child cognitive functioning will be assessed with a formal psychological test of cognitive functioning. According to age, the parents will complete a standardized behavioral and HRQoL questionnaire. Academic performance will be assessed by collecting the most recent CITO test scores from the Dutch Pupil monitoring system developed by the National Institute for Educational Measurement. Assessment of the prevalence of possible late effects of IVIg on the immune system will be assessed by questionnaires about the prevalence of allergies, astma, eczema and course of infections by questionnaires. Parents and children, when 12 years old or older, are asked for consent to request the medical letters from the maternity or neonatology ward to obtain perinatal and neonatal data.

No laboratory tests will be performed in this study, however data of the laboratory tests that were performed at timepoint of diagnosing FNAIT will be involved in this study.

After assessment a report will be made from the observations and test results, this report will be sent to the parents.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with FNAIT during pregnancy or postnatal, at moment of inclusion 2 to 16 years of age.
* Children living in the Netherlands.
* Parents or guardian aged ≥ 18 years old, with parental authority.
* Written informed consent form both parents with, form being approved by Ethic Committee.

Exclusion Criteria:

* Children born with congenital and/or chromosomal abnormalities.
* Children that passed away before inclusion.

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children born between 2002 and 2017 and diagnosed with FNAIT are eligible for this study. They will be invited for an assessment at our outpatient clinic. FNAIT cases that were not antenatally treated with IVIg will be eligible for the study (cohort 1), as well as FNAIT cases which were anticipated antenatally by materal IVIg administration (cohort 2).
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-12-17 (Estimated); Study Completion 2021-12-17 (Estimated)

PRIMARY OUTCOMES:
Cognitive test score | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  IQ test score calculated from a standardized cognitive test.

SECONDARY OUTCOMES:
Neurodevelopmental injury (NDI) | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  NDI is a composite outcome of:
  * Cerebral palsy ≥ grade II according to Gross Motor Classification System (GMFCS)
  * Impaired cognitive, language and/or motor development (test scores <70)
  * Bilateral blindness and/or bilateral deafness
  * Bilateral deafness requiring amplification
Health Related Quality of Life | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Health Related Quality of Life score calculated from the PedsQol questionnaire.
Cerebral Palsy | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Spastic bilateral, spastic unilateral or mixed Classification by European CP Network
Bilateral blindness | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Blind or partially sighted.
Bilateral deafness | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Needing hearing aids.
Behaviour test score | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Behaviour test score bases on Child Behavior Checklist
Abnormal course or incidence of infections | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Need to refer to an immunologist or the need to preform diagnostics based on history taking according to the Dutch guidelines.
Prevalence of eczema | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Number of children that suffer from eczema.
Prevalence of allergies | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Number of children that suffer from allergies
Patient reported anaphylaxis | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Serious allergic reaction, requiring urgent medical treatment with epinephrine.
Poor control of allergic rhinitis | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  CARAT score of upper airways < 8
Poor control of asthma | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  CARAT score of lower airways < 16.
Academic performance | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  The latest test scores from primary school will be requested. Three academic domains will be assessed; arithmetic and spelling performance and measurements on reading comprehension.

OTHER OUTCOMES:
Maternal characteristics | Measured at delivery of the child that is assessed. Calculated in years.
  Age mother at delivery
Obstetric history | Measured at delivery of the child that is assessed.
  History of pre-eclampsia, miscarriages or intra uterine fetal demise
Gravidity/Parity | Measured at delivery of the child that is assessed.
  Gravidity/Parity
Mode parturition | Measured at delivery of the child that is assessed.
  Mode parturition
Gestational age at birth | Measured at delivery of the child that is assessed. Gestational age expressed in days.
  Gestational age at birth in days
Birthweight | Measured at delivery of the child that is assessed, measurement directly after birth.
  Birthweight in grams
Apgar score | Measured at delivery of the child that is assessed, measured at 1, 5 and 10 minutes after birth.
  Apgar score
anti-HPA specificity | Measured at diagnosis of FNAIT, during pregnancy or until 1 week after birth.
  HPA specificity of the antibody found in the presence of an HPA incompatibility between mother and fetus.
Platelet count | Lowest platelet count measured between birth and 7 days after birth.
  Lowest platelet count
Platelet transfusion | Platelet transfusion between birth and 7 days after birth.
  Any platelet transfusion.
Neonatal IVIG treatment | Between birth and 7 days after birth.
  Any administration of IVIG after birth.
Skin bleeding manifestations | Between birth and 7 days after birth.
  Petechiae, purpura or hematoma diagnosed by the caretaker at neonatal period (gynecologist, pediatrician or midwife).
Intracranial hemorrhage | Between birth and 7 days after birth.
  Any intracranial hemorrhage
Convulsions | Between birth and 7 days after birth.
  Any paroxysmal, repetitive or stereotypical events interpreted as neonatal convulsions by a pediatrician.
Organ bleeding | Between birth and 7 days after birth.
  Bleeding in any organ located in the thorax or abdomen
Respiratory distress syndrome | Between birth and 7 days after birth.
  Requiring mechanical ventilation and/or surfactant.
Perinatal asphyxia | Diagnosed within 24 hours after birth.
  One of the following criteria; Apgar score < 7 and/or umbilical cord pH ≤ 7.0.
Proven early onset neonatal sepsis | Between birth and 7 days after birth.
  Positive blood culture within 72 hours postpartum and clinical suspicion of a neonatal sepsis.
Necrotizing enterocolitis | Between birth and 28 days after birth.
  Bells Stage 2 or higher.
Family history (first degree) of allergy, asthma or eczema | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Positive when 1st degree of family members receive daily treatment for asthma or eczema. Or when a family member wears an epinephrine pencil because of a severe allergy.
Ethnic origin of the parents | Asked at study enrollment.
  Ethnic origin of mother and father.
Parent smoking | Within 1 month before study enrollment.
  Any person living in the household of the child smoking one or more cigarettes a day.
Day-care visit | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  When child is in day care at least one day a week.
Educational level of the parents | From birth until study enrollment. Average age of the participants is expected to be 8 years old.
  Highest level of graduation of the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Lopriore, Prof. MD PhD, Principal Investigator — Department of Neonatology, Leiden University Medical Center; Masja de Haas, Prof. MD PhD, Principal Investigator — Stichting Sanquin Bloedvoorziening
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
In principle we do not share individual participant data with other researchers. If there is a request on sharing data this request is first submitted to the project leader (J.M.M. van Klink) or the principal investigators (E. Lopriore or M. de Haas). If they agree upon sharing data this request will be sent to the scientific committee of the Department of Pediatrics. If the project leader or scientific committees give permission for access to the data, the request is sent to a the METC of the LUMC. The METC will evaluate whether the purpose of reuse is in line with the informed consent.

REFERENCES:
- [Background] Dreyfus M, Kaplan C, Verdy E, Schlegel N, Durand-Zaleski I, Tchernia G. Frequency of immune thrombocytopenia in newborns: a prospective study. Immune Thrombocytopenia Working Group. Blood. 1997 Jun 15;89(12):4402-6. PMID 9192764
- [Background] Williamson LM, Hackett G, Rennie J, Palmer CR, Maciver C, Hadfield R, Hughes D, Jobson S, Ouwehand WH. The natural history of fetomaternal alloimmunization to the platelet-specific antigen HPA-1a (PlA1, Zwa) as determined by antenatal screening. Blood. 1998 Oct 1;92(7):2280-7. PMID 9746765
- [Background] Winkelhorst D, Kamphuis MM, Steggerda SJ, Rijken M, Oepkes D, Lopriore E, van Klink JMM. Perinatal Outcome and Long-Term Neurodevelopment after Intracranial Haemorrhage due to Fetal and Neonatal Alloimmune Thrombocytopenia. Fetal Diagn Ther. 2019;45(3):184-191. doi: 10.1159/000488280. Epub 2018 May 4. PMID 29730660
- [Background] Bussel JB, Berkowitz RL, Lynch L, Lesser ML, Paidas MJ, Huang CL, McFarland JG. Antenatal management of alloimmune thrombocytopenia with intravenous gamma-globulin: a randomized trial of the addition of low-dose steroid to intravenous gamma-globulin. Am J Obstet Gynecol. 1996 May;174(5):1414-23. doi: 10.1016/s0002-9378(96)70582-3. PMID 9065105
- [Background] Winkelhorst D, Murphy MF, Greinacher A, Shehata N, Bakchoul T, Massey E, Baker J, Lieberman L, Tanael S, Hume H, Arnold DM, Baidya S, Bertrand G, Bussel J, Kjaer M, Kaplan C, Kjeldsen-Kragh J, Oepkes D, Ryan G. Antenatal management in fetal and neonatal alloimmune thrombocytopenia: a systematic review. Blood. 2017 Mar 16;129(11):1538-1547. doi: 10.1182/blood-2016-10-739656. Epub 2017 Jan 27. PMID 28130210
- [Background] Ward MJ, Pauliny J, Lipper EG, Bussel JB. Long-term effects of fetal and neonatal alloimmune thrombocytopenia and its antenatal treatment on the medical and developmental outcomes of affected children. Am J Perinatol. 2006 Nov;23(8):487-92. doi: 10.1055/s-2006-954958. Epub 2006 Nov 8. PMID 17094038
- [Background] Radder CM, de Haan MJ, Brand A, Stoelhorst GM, Veen S, Kanhai HH. Follow up of children after antenatal treatment for alloimmune thrombocytopenia. Early Hum Dev. 2004 Oct;80(1):65-76. doi: 10.1016/j.earlhumdev.2004.05.007. PMID 15363839
- [Background] Yougbare I, Lang S, Yang H, Chen P, Zhao X, Tai WS, Zdravic D, Vadasz B, Li C, Piran S, Marshall A, Zhu G, Tiller H, Killie MK, Boyd S, Leong-Poi H, Wen XY, Skogen B, Adamson SL, Freedman J, Ni H. Maternal anti-platelet beta3 integrins impair angiogenesis and cause intracranial hemorrhage. J Clin Invest. 2015 Apr;125(4):1545-56. doi: 10.1172/JCI77820. Epub 2015 Mar 16. PMID 25774504
- [Background] van Gils JM, Stutterheim J, van Duijn TJ, Zwaginga JJ, Porcelijn L, de Haas M, Hordijk PL. HPA-1a alloantibodies reduce endothelial cell spreading and monolayer integrity. Mol Immunol. 2009 Jan;46(3):406-15. doi: 10.1016/j.molimm.2008.10.015. Epub 2008 Nov 26. PMID 19038456
- [Background] Tiller H, Kamphuis MM, Flodmark O, Papadogiannakis N, David AL, Sainio S, Koskinen S, Javela K, Wikman AT, Kekomaki R, Kanhai HH, Oepkes D, Husebekk A, Westgren M. Fetal intracranial haemorrhages caused by fetal and neonatal alloimmune thrombocytopenia: an observational cohort study of 43 cases from an international multicentre registry. BMJ Open. 2013 Mar 22;3(3):e002490. doi: 10.1136/bmjopen-2012-002490. PMID 23524102
- [Background] Janssen J, V.N., Engelen R, et al., Wetenschappelijke verantwoording van de toetsen LOVS rekenen-wiskunde voor groep 3 tot en met 8. [Scientific justification of the mathematics test for grade 1 until grade 6]. 2010, Cito: Arnhem.
- [Background] Mols A, K.F., Wetenschappelijke verantwoording van de toetsen Spelling nietwerkwoorden voor groep 7 en 8. [Scientific justification of the spelling test for grade 5 and 6]. . 2010, Cito: Arnhem.
- [Background] Weekers A, G.I., Kleintjes F, et al., Wetenschappelijke verantwoording papieren toetsen Begrijpend lezen voor groep 7 en 8. [Scientific justification of the reading comprehension test for grade 5 and 6]. 2011, Cito: Arnhem.
- [Background] Gilijns P, V.L., Het CITO leerlingvolgsysteem: Met het oog op de praktijk [The CITO pupil monitoring system: focus on practice]. Pedagogische Studiën 1992. 86:291-6.
- [Background] Touwen BC, Hempel MS, Westra LC. The development of crawling between 18 months and four years. Dev Med Child Neurol. 1992 May;34(5):410-6. doi: 10.1111/j.1469-8749.1992.tb11453.x. PMID 1592193
- [Background] Bayley, N., Bayley scales of infant and toddler development-Third edition. 2006: San Antonio, TX: Pearson Education, Inc.
- [Background] Wechsler, D., Wechsler Preschool and Primary Scale of Intelligence - Third Edition (WPPSI-III-NL). 2002: TX, The Psychological Corporation.
- [Background] Wechsler, D., Wechsler Intelligence Scale for Children (5th ed.). 2014a, San Antonio, TX: NCS Pearson
- [Background] Verhulst, F.C., J. van der Ende, and H.M. Koot,, Child Behavior Checklist (CBCL)/4-18 manual. 1996: Rotterdam: Afdeling Kinder- en Jeugdpsychiatrie, Sophia Kinderziekenhuis/Academisch Ziekenhuis Rotterdam/ Erasmus Universiteit Rotterdam.
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Emons JA, Flokstra BM, de Jong C, van der Molen T, Brand HK, Arends NJ, Amaral R, Fonseca JA, Gerth van Wijk R. Use of the Control of Allergic Rhinitis and Asthma Test (CARATkids) in children and adolescents: Validation in Dutch. Pediatr Allergy Immunol. 2017 Mar;28(2):185-190. doi: 10.1111/pai.12678. Epub 2016 Dec 23. PMID 27801950
- [Background] Driessen, G.J., Richtlijn diagnostiek naar onderliggende aandoeningen bij kinderen met recidiverende luchtweginfecties. 2016.
- [Background] Foundation, J.M. 10 Warning signs of primary immunodeficiency. 2016 [cited 2019 31-05].
- [Background] UNESCO, Institute for Statistics. International standard classification of education: ISCED 2011. 2012, UNESCO Institute for Statistics, : Montreal.
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Winkelhorst D, Oepkes D, Lopriore E. Fetal and neonatal alloimmune thrombocytopenia: evidence based antenatal and postnatal management strategies. Expert Rev Hematol. 2017 Aug;10(8):729-737. doi: 10.1080/17474086.2017.1346471. Epub 2017 Jun 29. PMID 28644735
- [Background] Volpe JJ. Intraventricular hemorrhage and brain injury in the premature infant. Diagnosis, prognosis, and prevention. Clin Perinatol. 1989 Jun;16(2):387-411. PMID 2663308
- [Background] Fonseca JA, Nogueira-Silva L, Morais-Almeida M, Azevedo L, Sa-Sousa A, Branco-Ferreira M, Fernandes L, Bousquet J. Validation of a questionnaire (CARAT10) to assess rhinitis and asthma in patients with asthma. Allergy. 2010 Aug;65(8):1042-8. doi: 10.1111/j.1398-9995.2009.02310.x. Epub 2010 Feb 1. PMID 20121755
- [Derived] de Vos TW, van Zagten M, de Haas M, Oepkes D, Tan RNGB, van der Schoot CE, Steggerda SJ, de Vries LS, Lopriore E, van Klink JMM. Children Newly Diagnosed with Fetal and Neonatal Alloimmune Thrombocytopenia: Neurodevelopmental Outcome at School Age. J Pediatr. 2023 Jul;258:113385. doi: 10.1016/j.jpeds.2023.02.031. Epub 2023 Mar 16. PMID 36933767

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT04529382/Prot_SAP_000.pdf